CLINICAL TRIAL: NCT04640753
Title: Peroral Endoscopic Myotomy for the Treatment of Achalasia: A Single-center Registry
Brief Title: Peroral Endoscopic Myotomy for the Treatment of Achalasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 031.GID.2018.D
Record Dates: First submitted 2019-11-27; First posted 2020-11-23 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic procedure for achalasia — POEM procedure will have a high technical feasibility, with effective clinical resolution of symptoms both in the short and long term.

SUMMARY:
There will be a retrospective chart review for patients who underwent endoscopic procedures and POEM from 06/2016 - 01/2019 & a prospective chart review will be performed for patients who will undergo endoscopic procedures and POEM from 02/2019 - 06/2021

DETAILED DESCRIPTION:
Subjects will undergo no additional tests and procedures as part of this study. All data will be collected from patient's electronic health records (EHR) of the hospital In addition; a prospective chart review will be performed for patients who will undergo endoscopic procedures and POEM from 02/2019 - 06/2021. All the subjects enrolled in prospective chart review will be first consented for their study participation. Subjects will undergo a clinically indicated endoscopic procedure and POEM and subsequent follow-up clinical visits as part of their standard medical care. All procedures, barring research activities such as consenting and data collection from Electronic Health Records, will be either clinically indicated and/or standard of care.

* Each patient in the study will be assigned a Case ID number to de-identify their personal health information during data collection
* The Case ID number connecting the patient to the personal health information will be in an encrypted electronic file on a computer that can only be accessed by study members at MDMC.
* A procedure report and outpatient clinical records for each subject's POEM procedure will be used to record each patient's data for the registry
* That data will only be shared by members of the study (PIs, research coordinator) who require it for conducting of data collection/interpretation

"Disclaimer: Any cost associated with the procedures stated herein will be billed directly to you or to your insurance (as applicable)."

ELIGIBILITY:
Inclusion Criteria:

* Any discharged patient who has undergone clinically indicated and/or standard of care POEM for the treatment of Achalasia from 6/2016 to 6/2021.
* Above or equal to 18 years of age

Exclusion Criteria:

* Any patient who has not undergone POEM for the treatment of Achalasia.
* Below 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There will be a retrospective chart review for patients who underwent endoscopic procedures and POEM from 06/2016 - 01/2019. In addition; a prospective chart review will be performed for patients who will undergo endoscopic procedures and POEM from 02/2019 - 06/2021.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-02-05 (Estimated)

PRIMARY OUTCOMES:
Decrease or no symptoms of chest pain | upto 180 days
  To continue and review our treatment outcomes, patient safety in cases with achalasia, we follow up after the procedure up to 180 days. Follow-up period varies from patient to patient.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided